CLINICAL TRIAL: NCT00970879
Title: Prevention of Pregnancy-associated Malaria in HIV-infected Women : Randomised Controlled Trial Testing Cotrimoxazole Prophylaxis Versus Intermittent Preventive Treatment With Mefloquine
Brief Title: Prevention of Pregnancy-associated Malaria in HIV-infected Women: Cotrimoxazole Prophylaxis Versus Mefloquine
Acronym: PACOME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Sidaction (Other); Saint Antoine University Hospital (Other); National University Hospital, Cotonou (Other); Université d'Abomey-Calavi (Other); Ministry of Health, Benin (Other Government)
Responsible Party: Principal Investigator, Lise Denoeud-Ndam, MD, MPH, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRD-Sidaction-01
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Malaria in Pregnancy; HIV Infections
Keywords: malaria; pregnancy; HIV; prevention; cotrimoxazole; mefloquine
MeSH Terms: conditions — HIV Infections; Malaria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cotrimoxazole (high) (Experimental): CD4 cell count≥350/mm3
  Interventions: Drug: cotrimoxazole
- mefloquine (Active Comparator): CD4 cell count≥350/mm3
  Interventions: Drug: mefloquine
- cotrimoxazole (low) (Experimental): CD4 cell count<350/mm3
  Interventions: Drug: cotrimoxazole
- mefloquine & cotrimoxazole (Active Comparator): CD4 cell count<350/mm3
  Interventions: Drug: cotrimoxazole; Drug: mefloquine

INTERVENTIONS:
Drug: cotrimoxazole — 800 mg sulfamethoxazole and 160 mg trimethoprim daily, from 28 weeks of gestation until delivery
  Arms: cotrimoxazole (high); cotrimoxazole (low); mefloquine & cotrimoxazole
Drug: mefloquine — mefloquine 15 mg/Kg three times, between 16 and 28 weeks, 24 and 32 weeks, then 28 and 36 weeks of pregnancy
  Arms: mefloquine; mefloquine & cotrimoxazole

SUMMARY:
The purpose of this study is to evaluate the efficacy of cotrimoxazole prophylaxis in prevention of malaria during pregnancy in HIV-infected women, compared to intermittent preventive treatment with mefloquine.

DETAILED DESCRIPTION:
Malaria infection during pregnancy can have adverse effects on both mother and fetus, including maternal anaemia and low birth weight which are responsible for mother and infant mortality. It is a particular problem for women in their first and second pregnancies and for women who are HIV-positive. Maternal HIV infection potentiates many of these adverse effects. In HIV-infected women, the World Health Organization (WHO) advocates the use of insecticide-treated bednets, and drugs : If the CD4 cell count is below 350/mm3 or the HIV disease is in WHO stage 2, 3 or 4, cotrimoxazole prophylaxis for the prevention of pneumocystosis and toxoplasmosis is indicated, that is assumed to also protect those women from malaria. Otherwise, they have to receive at least three doses of intermittent preventive treatment (IPT), most commonly with sulfadoxine-pyrimethamine (SP) given at the antenatal care visits. If IPT with SP has been a subject of many investigations, cotrimoxazole efficacy has never been assessed in prevention of malaria during pregnancy.

The investigators aim to evaluate the efficacy of cotrimoxazole prophylaxis in prevention of malaria during pregnancy in HIV-infected women. The investigators postulate that cotrimoxazole prophylaxis is not inferior to IPT in all women, unrelated to their CD4 cell count. In the control arm, the investigators will use mefloquine as IPT. The safety and efficacy of this drug have already been assessed in HIV-negative patients (NCT00274235).

A randomized controlled trial will be conducted in five hospitals in Benin. Pregnant women will be enrolled both in the Antenatal Care unit and in the Infectious Diseases unit of each setting. All women will receive insecticide-treated bednets at enrolment. Randomization will be stratified by hospital and CD4 cell count range. Women assigned to cotrimoxazole will receive cotrimoxazole prophylaxis daily during all the course of pregnancy. Women assigned to mefloquine IPT will receive mefloquine three times during pregnancy. Women randomised in this arm and having a low CD4 cell count or an advanced HIV disease will also receive cotrimoxazole prophylaxis in prevention of HIV/AIDS opportunistic infections. Drug efficacy will be judged on the prevalence of placental malaria at delivery.

This study will contribute to updating the recommendations concerning the prevention of malaria during pregnancy in HIV-infected women.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV seropositivity
* Permanent residency in the study catchment's area
* Confirmed pregnancy, gestational age< 28 weeks
* More than 18 years of age
* Karnofsky index ≥80
* Willingness to deliver at the hospital
* Written informed consent

Exclusion Criteria:

* History of allergy to study drugs : sulpha drugs, mefloquine, quinine
* History or presence of major illnesses : severe renal disease , severe hepatic disease, severe neuropsychiatric disease
* Mefloquine or halofantrine received within the 4 weeks prior to enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2009-12; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
proportion of placental malaria (presence of parasites in the placental blood smear at delivery) | delivery

SECONDARY OUTCOMES:
placental malaria mean parasite density at delivery | delivery
proportion of low birth weight infants (<2500 g) and mean birth weight | delivery
proportion of maternal anaemia (<11g/dl) and severe maternal anaemia (<8g/dl) at delivery and during pregnancy | course of pregnancy and delivery
cord blood malaria infection at delivery (infant parasitemia) | delivery
pre-term deliveries (< 37 weeks) | delivery
spontaneous abortions (early:<28 weeks, late: ≥28 weeks) and still births | course of pregnancy
congenital anomalies | first 6 months of life
safety profile of the two treatments: proportion and detailed description of adverse effects in each treatment arm | course of pregnancy (mother) anf first 6 months of life (infant)
Mother-to-child HIV transmission rate in each treatment arm | 2 months after breastfeeding cessation
To document the effect of cotrimoxazole in reducing infections in HIV-infected women, we will measure the incidence of bacterial and parasitic infections (other than malaria) during pregnancy | course of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Marcel D Zannou, Professor, Principal Investigator — Cotonou University Hospital & Faculté des Sciences de la Santé, Benin; Pierre-Marie Girard, Professor, Study Chair — Saint Antoine Hospital, Assistance Publique-Hôpitaux se Paris; Michel Cot, MD, PHD, Study Director — Institut de Recherche pour le Developpement
Locations (5):
- Benin (5):
  - Hôpital d'Instruction des Armées Camp Guézo, Cotonou
  - Hôpital de la Mère et de l'Enfant Lagune, Cotonou
  - Hôpital de zone de Suru Lere, Cotonou
  - Unviversity Hospital Hubert Koutoukou Maga, Cotonou
  - Clinique Louis Pasteur, Porto-Novo

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Duvignaud A, Denoeud-Ndam L, Akakpo J, Agossou KV, Afangnihoun A, Komongui DG, Atadokpede F, Dossou-Gbete L, Girard PM, Zannou DM, Cot M. Incidence of malaria-related fever and morbidity due to Plasmodium falciparum among HIV1-infected pregnant women: a prospective cohort study in South Benin. Malar J. 2014 Jul 4;13:255. doi: 10.1186/1475-2875-13-255. PMID 24996807